CLINICAL TRIAL: NCT05452772
Title: 5-HT2A Agonist Psilocybin in the Treatment of Tobacco Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Alabama at Birmingham (Other); New York University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00326148; U01DA052174 (NIH)
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation; Smoking; Cigarettes; Cigarette Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Smoking; Cigarette Smoking | interventions — Psilocybin; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Active Comparator): 30 mg in session 1 and either 30 mg or 40 mg in session 2, with sessions 1 week apart. Dosing will be based on participants' responses to the Mystical Experiences Questionnaire (MEQ30), taken at the end of their first session. Participants with a score ≥60% of the maximum on the MEQ30 will remain at a dose of 30 mg of psilocybin for the second session. Participants with an MEQ30 score below 60% will receive a dose of 40 mg for the second session.
  Interventions: Drug: Psilocybin
- Niacin (Active Comparator): 150 mg in session 1 and either 150 mg or 200 mg in session 2, with sessions 1 week apart. Dosing will be based on participants' responses to the Mystical Experiences Questionnaire (MEQ30), taken at the end of their first session. Participants with a score ≥60% of the maximum on the MEQ30 will remain at a dose of 150 mg niacin for the second session. Participants with an MEQ30 score below 60% will receive a dose of 200 mg niacin for the second session.
  Interventions: Drug: Niacin

INTERVENTIONS:
Drug: Psilocybin — Participants will received two psilocybin sessions, 1 week apart
  Other Names: Active Experimental Group
  Arms: Psilocybin
Drug: Niacin — Participants will received two niacin sessions, 1 week apart
  Other Names: Active Comparator Group
  Arms: Niacin

SUMMARY:
This is a multi-site, double-blind, randomized clinical trial of the 5-HT2A receptor agonist psilocybin for smoking cessation. Four sites with experience in conducting psilocybin research will be involved in this trial: Johns Hopkins University (JHU), the University of Alabama at Birmingham (UAB), and New York University (NYU). The proposed study will treat 66 participants (22 at each site), randomized to receive either: 1) oral psilocybin (30 mg in session 1 and either 30 mg or 40 mg in session 2); or 2) oral niacin (150 mg in session 1 and either 150 mg or 200 mg in session 2), with sessions 1 week apart.

DETAILED DESCRIPTION:
This is a multi-site, double-blind, randomized clinical trial of the 5-HT2A receptor agonist psilocybin for smoking cessation. The investigators previously conducted an open-label pilot trial (N = 15) of psilocybin paired with cognitive behavior therapy (CBT). Data showed a biologically-verified 7-day point-prevalence abstinence rate of 67% at 12 months and 60% at 2.5 years (continuous abstinence rates: 53% and 47%, respectively). The investigators are now conducting an open-label randomized comparative efficacy trial of psilocybin vs. nicotine patch, both in combination with CBT. Interim results (N = 44; 22 per group) show greater biologically-verified abstinence rates at 12 months for psilocybin: 7-day point-prevalence: 59% vs. 27%; continuous abstinence: 36% vs. 9%. Despite these promising findings, the investigators have yet to conduct a double-blind study of psilocybin for smoking cessation. Furthermore, previous psilocybin study samples have been largely White with higher socioeconomic status (SES). The current trial will address these issues across four sites with experience in conducting psilocybin research: Johns Hopkins, the University of Alabama at Birmingham (UAB), and New York University (NYU). A diverse sample with regard to ethno-racial identity and SES will be recruited at each site. The proposed double-blind study will treat 66 participants (22 at each site), randomized to receive either: 1) psilocybin; 30 mg in session 1 and either 30 or 40 mg in session 2, with sessions 1 week apart; or 2) niacin; 150 mg in session 1 and either 150 mg or 200 mg in session 2, with sessions 1 week apart. Niacin was selected because it has been used as an active placebo in two previous randomized therapeutic trials of psilocybin, and the FDA has informed the investigators that niacin is the FDA's preferred active placebo for psilocybin. CBT will be administered to both groups and will allow the investigators to test psilocybin's efficacy above and beyond an established treatment approach. Biochemically-confirmed 7-day point-prevalence abstinence will be assessed throughout for up to 12 months. The investigators hypothesize that psilocybin (compared to niacin) will cause increased biologically-confirmed 7-day point-prevalence abstinence at 12-month follow-up. Based on pilot data, the investigators will test cognitive/psychological mediators of treatment response. The investigators hypothesize that psilocybin will be associated with improved cognitive control and decreased anticipation of withdrawal relief (from smoking) 1 day after the target quit date, which will be associated with greater 7-day point-prevalence abstinence at 12- month follow-up. This trial will provide a rigorous test of efficacy in a diverse study sample, and test relevant mechanisms, for an innovative smoking cessation treatment showing potential for substantial efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older
* Be a daily smoker (minimum of 5 cigarettes/day on a typical day and breath CO of 6 or greater at screening) with multiple unsuccessful previous quit attempts, and report a continued desire to quit smoking
* Read, write, and speak English
* Agree to abstain from smoking for the psilocybin/niacin session from 1 hour before psilocybin/niacin administration until at least 8 hours afterward
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of psilocybin/niacin administration
* Be healthy as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis lab tests. See Exclusion Criteria below for specific ECG and specific blood test criteria

Exclusion Criteria:

* The use of e-cigarettes or tobacco products other than machine-manufactured combustible cigarettes (e.g., cigarillos) on more than 5 of the previous 30 days
* Women who are pregnant (positive pregnancy test) or nursing, or are not practicing an effective means of birth control
* Positive urine drug screen for illicit drugs (excluding cannabis)
* Positive urine breath test for alcohol. Participants with positive tests will be rescheduled
* For blood samples, the following lab values will be exclusionary: transaminases greater than x2 the upper limit of normal lab reference range, hemoglobin less than 11 g/d, and creatinine clearance < 40 ml/min using the Cockroft-Gault equation.
* For ECG screening: The ECG will be read by a cardiologist. Corrected heart rate (QTc) greater than 450 msec will be excluded.
* Patients who have baseline vital signs that exceed the following measurements will be excluded from participation: Systolic blood pressure (SBP) > 139 mmHG, diastolic blood pressure (DBP)> 89 mmHG, and heart rate of <=95 beats per minute (BPM). The investigators will perform serial heart rate monitoring with 3 total attempts. That is, heart rate must be <=95 bpm on one of these attempts to be included in the study.
* Currently taking on a regular basis (e.g., daily) antidepressants of any drug class, antipsychotics, or monoamine oxidase inhibitors (MAOIs), or serotonin-acting dietary supplements (e.g., 5-hydroxy- tryptophan, St. John's wort). Currently taking efavirenz, Acetaldehyde dehydrogenase inhibitors such as disulfiram (Antabuse), Alcohol dehydrogenase inhibitors, or uridine diphosphate glucuronosyltransferase 1-9 (UGT1A9) inhibitors or uridine diphosphate glucuronosyltransferase 1-10 (UGT1A10) inhibitors such as phenytoin, regorafenib, eltrombopag. For individuals who have intermittent or "as needed" use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose
* Current use of medications for smoking cessation (i.e., varenicline, nicotine replacement products, bupropion)
* Current neurological illnesses including, but not limited to, seizure disorders, frequent migraines or on prophylaxis, multiple sclerosis, movement disorders, history of significant head trauma (loss of consciousness > 24 hours), or central nervous system (CNS) tumor
* Recent (within the past 12 months) or an extensive history of psychedelic use (>20 lifetime uses)
* Current or past history of meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder. Current or past history within the last 5 years of meeting DSM-5 criteria for alcohol or drug use disorder (excluding caffeine and nicotine) or severe major depression
* Recent (past year) history of suicidal behavior or attempt or high-level current suicidal ideation assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
* Have a first- or second-degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I or II disorder
* Currently meets DSM-5 criteria for Dissociative Disorder, Anorexia Nervosa, Bulimia Nervosa, Major Depression, or Post-traumatic Stress Disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Potential Efficacy (Smoking Cessation) | 12 months
  Smoking cessation will be dichotomously coded 7-day point prevalence abstinence at 12-month follow-up. This binary outcome (abstinent versus non-abstinent) will be verified via three measures of recent smoking-(1) timeline follow-back (TLFB), a self-report calendar completed retrospectively by participants indicating the number of cigarettes smoked each day; (2) exhaled carbon monoxide (CO), an objective and biological measure of smoking over approximately the past 24 hours; and (3) urinary cotinine level, an additional biological and objective measure of nicotine exposure and allows for detection of smoking or other nicotine product use over the previous six days. Though these measures are not study outcomes individually, they will verify 7-day point prevalence abstinence at 12-month follow-up - the primary outcome. Specifically, 0 cigarettes reported on the TLFB, breath CO of ≤6 ppm, and urine cotinine levels of <200ng/mL will be considered smoking abstinence.

SECONDARY OUTCOMES:
Prolonged Abstinence | 12 months
  A secondary measure of abstinence will be prolonged abstinence, defined as no smoking at all after the target quit date, with the exception that smoking lapses during an initial 2-week grace period after the target quit date are not counted.
Cognitive control (Multi-Source Interference Task) at Screening (Visit 0) | Approximately 4 weeks prior to the target quit date
  The Multi-Source Interference Task is a measure of cognitive control that requires participants to inhibit a prepotent response when engaged in a voluntary task-based action. The Multi-Source Interference Task will be administered at screening - approximately 4 weeks prior to the first psilocybin / niacin session (i.e., 4 weeks prior to the target quit date), and again at Visits 5 and 6.
Cognitive control (Multi-Source Interference Task) at Visit 5 | Approximately 1 day after the target quit date
  The Multi-Source Interference Task is a measure of cognitive control that requires participants to inhibit a prepotent response when engaged in a voluntary task-based action. The Multi-Source Interference Task will be administered at Visit 5 - 1 day after the first psilocybin / niacin session (i.e., 1 day after the target quit date), and again at Visit 6.
Cognitive control (Multi-Source Interference Task) at Visit 6 | Approximately 2 days after the target quit date
  The Multi-Source Interference Task is a measure of cognitive control that requires participants to inhibit a prepotent response when engaged in a voluntary task-based action. The Multi-Source Interference Task will be administered at Visit 6, the day of the second psilocybin / niacin session (i.e., 2 days after the target quit date).
Smoking Urges (Questionnaire on Smoking Urges; Factor 2) at Screening | Approximately 4 weeks prior to the target quit date
  The Questionnaire on Smoking Urges is a multidimensional assessment of smoking craving with demonstrated sensitivity to smoking cessation. Participants will respond using a 7-point scale, where 1 = "Strongly Disagree", 4 = "Neither Agree nor Disagree", and 7 = "Strongly Agree". The scale consists of 10 items and scores can range from 10 - 70, with higher scores reflecting stronger urges to smoke.The Questionnaire on Smoking Urges will be administered at screening - approximately 4 weeks prior to the first psilocybin / niacin session (i.e., 4 weeks prior to the target quit date), and again at Visits 5 and 6.
Smoking Urges (Questionnaire on Smoking Urges; Factor 2) at Visit 5 | Approximately 1 day after the target quit date
  The Questionnaire on Smoking Urges is a multidimensional assessment of smoking craving with demonstrated sensitivity to smoking cessation. Participants will respond using a 7-point scale, where 1 = "Strongly Disagree", 4 = "Neither Agree nor Disagree", and 7 = "Strongly Agree". The scale consists of 10 items and scores can range from 10 - 70, with higher scores reflecting stronger urges to smoke. The Questionnaire on Smoking Urges will be administered at Visit 5 - 1 day after the first psilocybin / niacin session (i.e., 1 day after the target quit date), and again at Visit 6.
Smoking Urges (Questionnaire on Smoking Urges; Factor 2) at Visit 6 | Approximately 2 days after the target quit date
  The Questionnaire on Smoking Urges is a multidimensional assessment of smoking craving with demonstrated sensitivity to smoking cessation. Participants will respond using a 7-point scale, where 1 = "Strongly Disagree", 4 = "Neither Agree nor Disagree", and 7 = "Strongly Agree". The scale consists of 10 items and scores can range from 10 - 70, with higher scores reflecting stronger urges to smoke. The Questionnaire on Smoking Urges will be administered at Visit 6, the day of the second psilocybin / niacin session (i.e., 2 days after the target quit date).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Johnson, Ph.D, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - New York University, New York, New York

REFERENCES:
- [Background] Grob CS, Danforth AL, Chopra GS, Hagerty M, McKay CR, Halberstadt AL, Greer GR. Pilot study of psilocybin treatment for anxiety in patients with advanced-stage cancer. Arch Gen Psychiatry. 2011 Jan;68(1):71-8. doi: 10.1001/archgenpsychiatry.2010.116. Epub 2010 Sep 6. PMID 20819978
- [Background] Johnson MW, Garcia-Romeu A, Cosimano MP, Griffiths RR. Pilot study of the 5-HT2AR agonist psilocybin in the treatment of tobacco addiction. J Psychopharmacol. 2014 Nov;28(11):983-92. doi: 10.1177/0269881114548296. Epub 2014 Sep 11. PMID 25213996
- [Background] Johnson MW, Garcia-Romeu A, Griffiths RR. Long-term follow-up of psilocybin-facilitated smoking cessation. Am J Drug Alcohol Abuse. 2017 Jan;43(1):55-60. doi: 10.3109/00952990.2016.1170135. Epub 2016 Jul 21. PMID 27441452
- [Background] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164